CLINICAL TRIAL: NCT05665465
Title: Neurobehavioral Mechanisms Linking Childhood Adversity to Increased Risk for Smoking
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00110997; 1R01DA054972-01A1 (NIH)
Record Dates: First submitted 2022-12-12; First posted 2022-12-27 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Adverse Childhood Experiences; Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Intervention Model Description: All participants will sample the three doses of nicotine spray in a counter-balanced crossover design.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will be administered 2 nasal sprays with a combined nicotine content of 0mg nicotine, 0.1mL
  Interventions: Drug: Placebo
- 0.5mg nicotine (Experimental): Participants will be administered 2 nasal sprays with a combined nicotine content of 0.5 mg nicotine, 0.1mL
  Interventions: Drug: Nicotine nasal spray 0.5 mg; Drug: Placebo
- 1mg nicotine (Experimental): Participants will be administered 2 nasal sprays with a combined nicotine content of 1.0 mg nicotine, 0.1mL
  Interventions: Drug: Nicotine nasal spray 0.5 mg

INTERVENTIONS:
Drug: Nicotine nasal spray 0.5 mg — Participants will be administered nicotine nasal spray and provide subjective reactions
  Other Names: Nicotrol
  Arms: 0.5mg nicotine; 1mg nicotine
Drug: Placebo — Participants will be administered placebo nasal spray and provide subjective reactions
  Arms: 0.5mg nicotine; Placebo

SUMMARY:
The purpose of this study is to evaluate how certain childhood experiences influences brain function and responses to nicotine exposure in a group of nonsmoking young adults. The investigators assess responses to nicotine exposure by giving participants a small amount of nicotine or placebo, and then asking them to answer questionnaires. The investigational drugs used in this study are a nicotine nasal spray (i.e., Nicotrol) and/or a nasal spray placebo (made of common kitchen ingredients, including a very tiny amount of pepper extract also called capsaicin). The investigators assess brain function through function magnetic resonance imaging (fMRI), which is a noninvasive procedure that uses a magnetic field to take pictures of your brain while you are performing certain tasks. This study will help us to learn more about why some childhood experiences (adverse childhood experiences, or ACEs) contribute to increased risk for smoking and other substance use.

DETAILED DESCRIPTION:
Individuals with a history of adverse childhood experiences (ACEs) are more likely to smoke cigarettes than those without, but little is known about the factors that account for this increased risk. This study will examine brain function in regions related to reward processing and inhibitory control, along with reactions to initial nicotine exposure to help explain why ACEs lead to increased risk for smoking. In this study, young adult non-smokers ages 18-21 (n=150) with a history of exposure to ACEs ranging from 0 to 4 or more will be enrolled to attend 7 visits including an MRI scan and administration of a nicotine nasal spray. Participants will complete an in-person screening visit, followed by a training visit to provide training for the MRI tasks and to acclimate them to the mock MRI scanner. They will then complete a functional neuroimaging scanning session to examine brain reactivity during a monetary reward task, an inhibitory control task, and during rest. Participants will then attend 3 separate visits in which subjective reactions to a nasal spray containing 0, .5, or 1 mg doses of nicotine will be measured. During a final choice session participants will choose to self-administer nicotine or placebo nasal spray. Breath and urine samples will be collected at each visit to test for recent smoking, alcohol use, or illicit drug use. Plasma samples will be collected at each fixed-dose session to assess nicotine and cotinine levels. All nicotine administration will occur during laboratory sessions, and the study physician will be on site or on call during all visits.

ELIGIBILITY:
Inclusion Criteria:

1. generally healthy
2. 18-21 years of age
3. never smoked a full cigarette or used an equivalent amount of other nicotine or tobacco products
4. no tobacco exposure in the past 3 years
5. expired air CO level ≤ 3 ppm
6. corroboration of non-smoking status from 2 collateral reporters
7. breath alcohol value = 0.000

Exclusion Criteria:

1. use of illegal drugs as measured by urine drug screen
2. reported history of illicit drug use > 10 times lifetime
3. lifetime history of alcohol use disorder
4. binge drinking > 5 times per month over the past 3 months
5. history of serious mental illness including bipolar or psychotic disorders
6. significant medical or unstable psychiatric disorders
7. systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg
8. heart rate ≥ 100 bpm
9. use of psychoactive medications (e.g., antidepressants, opioid analgesics, etc.) in the past 6 months
10. presence of conditions that would make fMRI unsafe (e.g., pacemaker)
11. brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder)
12. history of serious traumatic brain injury
13. claustrophobia
14. lack of firm resolve to refrain from cigarette, e-cigarette or other tobacco use in the coming year
15. pregnant, trying to become pregnant, or breastfeeding
16. inability to understand written and/or spoken English language
17. inability to attend all experimental sessions

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Subjective effects of nicotine nasal spray as measured by the Nicotine Effects Questionnaire | during fixed dose session, approximately 3 hrs
  subjective effects will be measured by the Nicotine Effects Questionnaire at the end of each fixed dose session. This scale measure positive reactions, negative reactions, and dizziness on a scale from 0-3 where 0 is none and 3 is intense.
Subjective effects of nicotine nasal spray as measured by a visual analog scale | during fixed dose session, approximately 3 hrs
  subjective effects will be measured on a visual analog scale at the end of each fixed dose session. Ratings will be provided on a scale of 0=not at all to 100=an awful lot.
Reinforcing effects of nicotine nasal spray | during choice session, approximately 4 hrs
  reinforcing effects will be measured by the number of choices for nicotine spray (range 0-8) during the forced choice session.
Percent BOLD signal change in ventral striatum | baseline, prior to intervention
  Percent blood oxygen level-dependent (BOLD) signal change during anticipation of monetary gain versus baseline during the Reward Guessing Task will be extracted from the bilateral ventral striatum
Percent BOLD signal change in inferior frontal gyrus | baseline, prior to intervention
  Percent BOLD signal change during "rare go" versus "no-go" trials during the Go/No-Go Task will be extracted from the right inferior frontal gyrus

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Sweitzer, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No